CLINICAL TRIAL: NCT06351267
Title: Combined Effects of Core Stability Exercises and Back Strengthening Exercises on Pregnancy-Induced Back Pain, Disability and Function.
Brief Title: Combined Effects of Core Stability Exercises and Back Strengthening Exercises on Pregnancy-Induced Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0568
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Stability Exercises and Back Strengthening exercises group: (Experimental): we will ask the patient to perform a combined exercise program of core stability exercises program with a back strengthening exercises program. 5 sessions per week and post-intervention assessment after 4 weeks follow-up
  Interventions: Other: Core Stability Exercises; Other: Back Strengthening exercises
- Core Stability Exercise group (Active Comparator): In this group, patients will only perform the Core Stability Exercises program. 5 sessions per week and post-intervention assessment after 4 weeks follow-up
  Interventions: Other: Core Stability Exercises

INTERVENTIONS:
Other: Core Stability Exercises — Core stability exercises will be used to strengthen the core muscles, which includes sets of exercises like pelvic tilts, wall squatting, bridging, bird dog and heel walking which targets core muscles.
Other: Back Strengthening exercises — Back strengthening exercises will be used to strengthen the back muscles which include sets of exercises that target back muscles like cat-cow exercise, child pose, heel sits, and kegels.
  Arms: Core Stability Exercises and Back Strengthening exercises group:

SUMMARY:
The study will be a Randomized controlled trial to check the combined effects of Core Stability Exercises with and without Back strengthening exercises in females with pregnancy-induced back pain, disability, and function so that we can examine the effect of the above techniques on pain, disability and function in pregnant females Non-probability convenience sampling technique will be used, subject following eligibility criteria from Society Hospital Nabipura Lahore will be randomly allocated in two groups. Group A participants will be given core stability exercises with back strengthening exercises, Group B participants will be given core stability exercises for 4 weeks. Assessment will be done via, Numeric Pain Rating Scale, Oswestry disability index questionnaire and Back pain Functional Scale.

DETAILED DESCRIPTION:
Pregnancy-inducedBack pain causes weakness of abdominal muscles and pelvic muscles which affects core stability and back strength of pregnant women. In this study, the effects of Core Stability Exercises with and without Back strengthening exercises in pregnancy-induced back pain population will be analyzed. This study will be a randomized controlled trial. Core stability exercises and Strengthening exercises program would be applied to pregnant females with pregnancy-induced back pain. Subjects meeting the predetermined inclusion criteria will be divided into two groups. Assessment will be done using the Numeric Pain Rating Scale (NPRS), Oswestry Disability Index Questionnaire, and Back Pain Functional Scale (BPFS). Subjects in one group will be treated with core stability exercises with back strengthening exercises, and the other will be treated with core stability exercises only. Each subject will receive a total of 20 treatment sessions, with 05 treatment sessions per week. Measurements will be recorded at the start and end of the treatment session. Recorded values will be analyzed for any change using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females
* Pregnant female in their second and third trimester.
* Multi gravida patient
* Low back pain intensity greater than 4 out of 10 on NPRS, indicating moderate to severe.

Exclusion Criteria:

* Placenta previa
* Bleeding or spotting
* Low back pain before pregnancy
* Pregnancy-induced hypertension
* Pudendal nerve entrapment syndrome.
* Not simultaneously partaking in pelvic floor physical therapy.
* No evoked tenderness upon palpation of levatorani sling at examination.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | up to 4 weeks
  The NPRS is a segmented numeric scale in which the respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. NPRS is anchored by terms describing pain severity extremes. changes from Baseline to 4 week
Oswestry Disability Index Questionnaire | up to 4 weeks
  The Oswestry disability index questionnaire gives subjective percentage score of level of function(disability) in activities of daily living in those rehabilitating from low back pain with level of disability in 10 everyday activities. Each item consists of 6 options with score 0-5. With 0 indicating least disability and 5 greater then total score will be calculated as percentage. 0% indicating no disability and 100% highest level of disability.
Back Pain Functional Scale (BPFS): | up to 4 weeks
  The BPFS is a subjective scale used to measure the patient physical function after low back pain. It consists of 12 items and total score of 60. The maximum score indicates maximum physical abilities of patient. 0 being no physical abilities and 60 being no difficulty in any activity

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Shafiq Dar, MS*, Principal Investigator — Riphah International University, Lahore, Pakistan
Locations (1):
- Society Hospital Nabipura, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kluge J, Hall D, Louw Q, Theron G, Grove D. Specific exercises to treat pregnancy-related low back pain in a South African population. Int J Gynaecol Obstet. 2011 Jun;113(3):187-91. doi: 10.1016/j.ijgo.2010.10.030. Epub 2011 Apr 1. PMID 21458811
- [Background] Ghaderi F, Mohammadi K, Amir Sasan R, Niko Kheslat S, Oskouei AE. Effects of Stabilization Exercises Focusing on Pelvic Floor Muscles on Low Back Pain and Urinary Incontinence in Women. Urology. 2016 Jul;93:50-4. doi: 10.1016/j.urology.2016.03.034. Epub 2016 Apr 5. PMID 27059833
- [Background] Weis CA, Nash J, Triano JJ, Barrett J. Ultrasound Assessment of Abdominal Muscle Thickness in Women With and Without Low Back Pain During Pregnancy. J Manipulative Physiol Ther. 2017 May;40(4):230-235. doi: 10.1016/j.jmpt.2017.02.002. Epub 2017 Apr 12. PMID 28410762
- [Background] Richardson CA, Jull GA. Muscle control-pain control. What exercises would you prescribe? Man Ther. 1995 Nov;1(1):2-10. doi: 10.1054/math.1995.0243. PMID 11327788
- [Background] Mamipour H, Farazmehr S, Negahban H, Nazary-Moghadam S, Dehghan-Manshadi F, Navi Nezhad M, Jafari S, Sharifzadeh M. Effect of Core Stabilization Exercises on Pain, Functional Disability, and Quality of Life in Pregnant Women With Lumbar and Pelvic Girdle Pain: A Randomized Controlled Trial. J Manipulative Physiol Ther. 2023 Jan;46(1):27-36. doi: 10.1016/j.jmpt.2023.05.005. Epub 2023 Jul 7. PMID 37422748
- [Background] Katonis P, Kampouroglou A, Aggelopoulos A, Kakavelakis K, Lykoudis S, Makrigiannakis A, Alpantaki K. Pregnancy-related low back pain. Hippokratia. 2011 Jul;15(3):205-10. PMID 22435016
- [Background] Barbier M, Blanc J, Faust C, Baumstarck K, Ranque-Garnier S, Bretelle F. Standardized Stretching Postural postures to treat low-back pain in pregnancy: the GEMALODO randomized clinical trial. Am J Obstet Gynecol MFM. 2023 Oct;5(10):101087. doi: 10.1016/j.ajogmf.2023.101087. Epub 2023 Jul 11. PMID 37437692